CLINICAL TRIAL: NCT05398523
Title: Association of Frailty, Balance, and Depression With Activities of Daily Living in Older Adults
Brief Title: Activities of Daily Living in Older Adults
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Seda Saka, PT PhD, Halic University
Other Study IDs: ssaka5
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Geriatrics
Keywords: Frailty; balance; depression; activities of daily living
MeSH Terms: conditions — Frailty; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to maintain independence and prevent disability, it is essential to identify associated factors and reduce functional loss due to concomitant diseases. This study aimed to examine the effects of frailty, balance, and depression on the performance of activities of daily living in older adults. All participants were assessed using the Mini Mental State Test, simple FRAIL scale, Geriatric Depression Scale-Short Form, and Lawton Instrumental Activities of Daily Living Scale (IADL).

DETAILED DESCRIPTION:
As the global population becomes older, the importance of preserving health, function, and quality of life is being increasingly recognized. In order to maintain independence and prevent disability, it is essential to identify associated factors and reduce functional loss due to concomitant diseases. This study aimed to examine the effects of frailty, balance, and depression on the performance of activities of daily living in older adults. All participants were assessed using the Mini Mental State Test, simple FRAIL scale, Geriatric Depression Scale-Short Form, and Lawton Instrumental Activities of Daily Living Scale (IADL).

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or older
* being able to understand and answer the questionnaires used for data collection
* having mental competency as demonstrated by a score higher than 20 on the Mini Mental State Test

Exclusion Criteria:

* limited ambulation
* psychological problems

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: adults aged 65 years or older who were registered at Community Health Center No.1 in City Central Amasya.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2020-09-27 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Test | at the enrollment
  Cognitive function was assessed using the MMST, which consists of 11 items. The MMST has a maximum score of 30 points; scores above 24 points are considered sufficient and scores lower than 20 indicate cognitive impairment

SECONDARY OUTCOMES:
FRAIL scale | at the enrollment
  This 5-item scale was developed by Morley et al. in 2012. People with a score of 0 points are regarded as normal, 1-2 points as pre-frail, and 3-5 points as frail
Berg Balance Scale | at the enrollment
  Balance was assessed using the BBS, which was developed to measure balance performance. It includes 14 instructions, each of which is scored between 0-4 based on performance of the instruction. The BBS is administered in 10-20 minutes and the maximum score is 56. A score of 0-20 points indicates impaired balance, 21-40 points indicates acceptable balance, and 41-56 points indicates good balance
Geriatric Depression Scale-Short Form | at the enrollment
  The GDS-SF was used to assess the participants' depression level. The scale consists of 15 yes/no questions about the participant's feelings in the past week. Each item is scored 0 or 1, with a higher score indicating the presence of more depressive symptoms
Lawton Instrumental Activities of Daily Living Scale | at the enrollment
  The scale consists of 8 items including information about using the telephone, preparing food, shopping, doing daily household chores, doing laundry, using transport, using drugs, and managing money. Scores range from 0 (dependent) to 8 (independent)

CONTACTS AND LOCATIONS:
Overall Officials: Seda Saka, PT, PhD, Study Director — Haliç University
Locations (1):
- Haliç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vieira ER, Da Silva RA, Severi MT, Barbosa AC, Amick Iii BC, Zevallos JC, Martinez IL, Chaves PHM. Balance and Gait of Frail, Pre-Frail, and Robust Older Hispanics. Geriatrics (Basel). 2018 Jul 18;3(3):42. doi: 10.3390/geriatrics3030042. PMID 31011080
- [Result] Marques LT, Rodrigues NC, Angeluni EO, Dos Santos Pessanha FPA, da Cruz Alves NM, Freire Junior RC, Ferriolli E, de Abreu DCC. Balance Evaluation of Prefrail and Frail Community-Dwelling Older Adults. J Geriatr Phys Ther. 2019 Jul/Sep;42(3):176-182. doi: 10.1519/JPT.0000000000000147. PMID 28914718